CLINICAL TRIAL: NCT04552639
Title: A Randomized Control Trial Study Evaluating a Compulsive Exercise Group for Adolescent Inpatients With Eating Disorders
Brief Title: Evaluation of Compulsive Exercise Group Therapy for Eating Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newbridge House (Other)
Responsible Party: Principal Investigator, Gurdeep Aulakh, Assistant Psychologist, Newbridge House
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 281456
Record Dates: First submitted 2020-08-21; First posted 2020-09-17 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Eating Disorders in Adolescence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: There is an external statistician who will assess the outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (Active Comparator): Treatment as usual is offered. This includes; individual therapy, group therapy, dietetic support, occupational therapy, nursing and psychiatry, excluding the NEAT group.
  Interventions: Behavioral: Newbridge House treatment as usual
- Treatment as usual and NEAT group (Experimental): Treatment as usual is offered. This includes; individual therapy, group therapy, dietetic support, occupational therapy, nursing and psychiatry, alongside NEAT group.
  Interventions: Behavioral: Newbridge Eating disorders Activity Treatment group

INTERVENTIONS:
Behavioral: Newbridge Eating disorders Activity Treatment group — A compulsive exercise cognitive-behavioural based group, for children and adolescents diagnosed with an eating disorder. It was devised for eating disorders including Anorexia Nervosa, Bulimia Nervosa and Other Specified Feeding or Eating Disorder. This treatment is semi-structured and problem-oriented, which focuses on tackling the factors and processes that maintain compulsive exercise behaviour.
  Arms: Treatment as usual and NEAT group
Behavioral: Newbridge House treatment as usual — Multi-disciplinary eating disorder treatment (including; psychiatry, individual therapy, group therapy, dietetic support, occupation therapy and nursing excluding NEAT group).
  Arms: Treatment as usual

SUMMARY:
The study aims to generate hypotheses about whether a group intervention is effective in reducing motivation to compulsive exercise and/or eating disorder psychopathology when compared with a control group. This will be explored through a Randomized Control Trial.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients at Newbridge House
* Aged 11-18
* Primary diagnosis of any form of eating disorder
* Females

Exclusion Criteria:

* Previously received NEAT group at Newbridge House
* Aged under 10 years
* Severe learning disability
* Inpatients without compulsive exercise behaviours
* Day patients
* Co-morbid psychosis
* Males

Ages: 11 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Compulsive Exercise Test | Week 1 and week 7

SECONDARY OUTCOMES:
Change in Eating Disorder Examination Questionnaire | Week 1 and week 7

CONTACTS AND LOCATIONS:
Locations (1):
- Newbridge House, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No